**Informed Consent for Research** 

Clinical Interventions template - Version: March 30, 2018

IRB Protocol Number: PRO00027931

IRB Approval Period: 9/25/2018 - 2/26/2019

**EFFECTIVE** 

9/25/2018

MCW/FH IRB

# Medical College of Wisconsin and Froedtert Hospital INTRODUCTION TO THE INFORMED CONSENT

| Name of Subject: |
|------------------|

Induction of Remission and Response of Vedolizumab Monotherapy Vs. Combination Therapy with Tacrolimus in Patients with Moderately to Severely Active Ulcerative Colitis

Andres Yarur, MD
Department of Medicine / Gastroenterology
414-955-6729
Medical College of Wisconsin
8701 Watertown Plank Road
Milwaukee WI 53226

You are invited to take part in this research. You can decide whether to take part in this project or not. You are free to say yes or no. If there is anything that you do not understand, please ask questions.

## **Definitions**

**Ulcerative Colitis** – a type of chronic inflammatory bowel disease (IBD) characterized by inflammation, deterioration/narrowing of the intestinal wall, and/or the presence of ulcers in the colon. Some common symptoms are stool urgency, abdominal pain, blood in the stool, and constipation.

**Vedolizumab** – a drug used for the management and treatment of inflammatory bowel disease (Entyvio)

**Tacrolimus** – a drug used for suppressing the immune system in patients that have had organ transplants (Prograf). It is not approved by the FDA for the treatment of IBD.

**Standard of Care** – Routine care; care you would receive to treat your IBD regardless of study participation.

**Flexible Sigmoidoscopy –** an examination that looks at the inside of the lower or sigmoid portion of the colon (large intestine) and rectum

**Biopsy** – tissue samples, about the size of a pencil tip, snipped from the bowel during the sigmoidoscopy procedure.

**Informed Consent for Research** 


IRB Protocol Number: PRO00027931

IRB Approval Period: 9/25/2018 - 2/26/2019

## **EFFECTIVE**

9/25/2018

MCW/FH IRB

#### **Purpose**

This project is being done to find out whether a new combination of drugs for ulcerative colitis, vedolizumab with tacrolimus, is better than vedolizumab alone.

#### Length

 You will be in this research project for about 32 weeks.

## **Procedures**

## List of visits:

Screening

- Total Number: 1

- Total Time: up to 8 hours

Baseline Visit

Total Number: 1Total Time: 2 hours

Weeks 2,6,8,14

Total Number: 4Total Time: 1.5 hours

Lab visits (blood draws)/phone calls

Total Number: up to 36Total Time: varies

Week 30 phone call

- Total Number: 1

- Total Time: 20 minutes

# Procedures that will occur at various visits:

## **Invasive Procedures**

 During screening and at week 6, you will have a flexible sigmoidoscopy.
 At each visit, and sometimes between visits, you will have your blood drawn for labs.

## Non-invasive Procedures

 You will be asked to provide a stool sample 3 times.

## Risks

This is a brief list of the most commonly seen side effects. The *full consent form* after this introduction contains a more complete list of potential research risks.

## Drug risks:

- Kidney injury
- Tremor
- Infection

## Flexible Sigmoidoscopy risks:

 Heavy or ongoing bleeding from biopsy, pain, bloating, perforation, nausea, vomiting, irritation

**Informed Consent for Research** 


IRB Protocol Number: PRO00027931

IRB Approval Period: 9/25/2018 - 2/26/2019

**EFFECTIVE** 

9/25/2018

MCW/FH IRB

## **Benefits**

We don't know if this project will help you. Your condition may get better but it could stay the same or even get worse.

## My Other Options

You do not have to join this project. Your other options may include:

- Joining a different project
- Routine care for this condition
- Getting no treatment for this condition

If you have more questions about this project at any time, you can call Dr. Yarur at 414-955-6858

If you have questions about your rights as a participant, want to report any problems or complaints, or offer input, you can call the MCW/Froedtert Hospital Research Subject Advocate at 414-955-8844.

**Informed Consent for Research** 


IRB Protocol Number: PRO00027931

IRB Approval Period: 9/25/2018 - 2/26/2019

**EFFECTIVE** 

9/25/2018

MCW/FH IRB

#### **CONSENT TO PARTICIPATE IN RESEARCH**

#### A1. INTRODUCTION - WHY ARE WE ASKING YOU TO PARTICIPATE?

You are being invited to participate in this research because you have moderate to severe ulcerative colitis and are starting vedolizumab as part of your clinical care. Because of your condition, you may be eligible for a research project on a new drug for ulcerative colitis, to be used with your vedolizumab.

A total of about 20 people are expected to participate in this research, all at the Medical College of Wisconsin/Froedtert Hospital.

The Director of the project is Dr. Andres Yarur in the Department of Medicine / Gastroenterology. A research team works with Dr. Yarur. You can ask who these people are.

Takeda, a drug company, is funding the research.

## **A2. DO I HAVE TO PARTICIPATE?**

You can decide whether to take part in this research or not. You are free to say yes or no. If you say no, your regular medical care will not change. Even if you join this project, you do not have to stay in it. You may stop at any time.

A research project is different from routine medical care in three ways: 1) there are extra risks that we will tell you about in this form; 2) you may have some extra medical tests and visits; 3) the research procedures, tests and visits follow a set plan that must be kept.

## A3. WHY IS THIS PROJECT BEING DONE?

In this study we want to find out whether a new combination of drugs for ulcerative colitis, vedolizumab with tacrolimus, is better than vedolizumab alone. Vedolizumab is an FDA-approved treatment for ulcerative colitis. To do this, we will compare the two treatments in people with ulcerative colitis and see which one reduces symptoms faster or better, and which one is safer (causes fewer problems). Tacrolimus is approved by the U.S. Food and Drug Administration for use in patients, but not for treating patients with ulcerative colitis. The combination of vedolizumab with tacrolimus may have advantages over vedolizumab alone, but we won't know until we do more research.

We don't know if this study will help you. Your condition may get better but it could stay the same or even get worse. We hope the information from this study will help us develop a better treatment for ulcerative colitis in the future.

**Informed Consent for Research** 


IRB Protocol Number: PRO00027931

IRB Approval Period: 9/25/2018 - 2/26/2019

**EFFECTIVE** 

9/25/2018

MCW/FH IRB

#### **B1. WHAT WILL HAPPEN IF I PARTICIPATE?**

At the end of this form, a table is attached. This table is the schedule of study procedures. Procedures that are done only for the study (research only) are highlighted. The other procedures are part of your standard of care or information pulled from your medical record.

## **Screening procedures:**

If you decide to join the study, some screening tests will be done first to see if you are eligible.

- You will be asked to sign this informed consent
- You will have a flexible sigmoidoscopy to determine the severity of your disease. Part of this procedure will include a biopsy for the lab to rule out an infection called CMV.

A flexible sigmoidoscopy is an examination that looks at the inside of the lower or sigmoid portion of the colon (large intestine) and rectum. The examination uses a tool called a colonoscope or flexible sigmoidoscope. On the day of the examination you may be given medicine prior to the examination to help you relax; you could have some discomfort during the examination. You will lie on your left side with your knees drawn up toward your chest. The colonoscope or flexible sigmoidoscope is inserted into the anus and, under visual control, is gently moved into the rectum and through the sigmoid colon. Air will be inserted through the scope to provide a better view and suction may be used to remove fluid or stool. You may feel pressure as the scope moves inside. Following the examination, you will be kept in an observation area for an hour or so until the effects of the medications (if administered) that have been given adequately wear off. Passing gas is necessary and should be expected. Feeling bloated and swollen are also common due to the air inflated into the bowel; this usually lasts only 30 to 60 minutes. You must plan to have someone take you home after the test, because you will be drowsy and unable to drive in the event sedating medication was administered. During the examination the study doctor looks at the lining of the bowel and snips tissue samples, called biopsies from the bowel for further study, to make sure you don't have an infection called CMV. Each biopsy is about the size of a pencil-tip.

- We will review some information from your medical record results of recent colonoscopy/sigmoidoscopy, labs, medications, and medical history relating to your ulcerative colitis
- A urine pregnancy test will be performed if you are a woman of child bearing potential.

If the screening information shows that you meet the requirements, then you will be able to start the study. If the screening information shows that you cannot be in the research study, the study doctors will discuss other options with you and/or refer you back to your regular doctor.

#### Research groups

To find out if vedolizumab with tacrolimus treats ulcerative colitis more effectively than vedolizumab alone, one group of people in the study will be given vedolizumab and tacrolimus, and a second group of people will be given vedolizumab and a placebo.

You should know that the placebo is a pill that contains no real medicine and we do not expect it will do anything for your health.

#### **Informed Consent for Research**


IRB Protocol Number: PRO00027931

IRB Approval Period: 9/25/2018 - 2/26/2019

#### **EFFECTIVE**

9/25/2018

MCW/FH IRB

Because no one knows which of the treatments is best, you will be randomized into one of the two study groups. One group will receive vedolizumab and tacrolimus, and one group will receive vedolizumab and a placebo. Randomization means that you are put into a group by chance. It is like flipping a coin. You will have an equal chance of being placed in either group.

Since the expectations of patients and doctors can influence the results of a study, neither you nor your study doctor can know which drug you will get until the study is over. This is called a blinded study. A computer program chooses which group you are in, and the pills in each group will look the same. In an emergency, your doctor can find out which drug you are taking.

# **Summary of Procedures:**

## **Baseline assessment**

- collect information from your routine care appointment, including vital signs, lab results, and scores for assessing the severity of your symptoms.
- begin study medication
- laboratory tests (phosphorus, magnesium, tacrolimus level)
   A stool sample is needed to measure fecal calprotectin. these are not part of your routine care and are considered research only

Weeks 2 and 8 - this visit is not part of your routine care and is considered research only

- vital signs (blood pressure, heart rate, temperature, weight)
- we will ask you about medications you are taking
- we will ask you about side effects you may be having
- laboratory tests (complete blood count [CBC], comprehensive metabolic panel, phosphorus and magnesium levels, tacrolimus level (these tests will require the collection of about 30 ml (2 tablespoons) of blood), pregnancy testing (at week 2 only)
- you will be asked to complete questionnaires/scores for assessing the severity of your symptoms

**Weeks 6 and 14** – these visits are part of your routine care, and only noted laboratory tests are considered to be for the study only

- vital signs (blood pressure, heart rate, temperature, weight)
- we will ask you about medications you are taking
- we will ask you about adverse events (side effects) you may be having
- flexible sigmoidoscopy (week 6 only)
- laboratory tests (CBC, CMP, CRP)
- tacrolimus, phosphorus, and magnesium levels, and a stool sample for fecal calprotectin – these are not part of your routine care and are considered research only
- pregnancy testing this is not part of your routine care and is considered research only
- you will be asked to complete questionnaires/scores for assessing the severity of your symptoms

## **Weekly Phone Call**

 The study coordinator will call you weekly for the first 14 weeks of the study to assess for side effects or concerns. At Week 12, your call will also include a reminder to stop your study medication.

#### **Informed Consent for Research**


IRB Protocol Number: PRO00027931

IRB Approval Period: 9/25/2018 - 2/26/2019

**EFFECTIVE** 

9/25/2018

MCW/FH IRB

#### Week 30

- review of your medical record
- phone call to ask you about your health and check for adverse events

You will also be asked to record your daily symptoms (stool frequency and rectal bleeding) in a diary for the 12 weeks that you are receiving the study drugs. This diary will be shared with the research team.

You will receive intravenous vedolizumab at Weeks 0 (baseline visit), 2, and 6, and every 8 weeks thereafter. This is part of your standard of care.

Tacrolimus (or placebo) will be started on the same day as your first vedolizumab dose. The tacrolimus/placebo is a tablet that you will take daily at home. The dose of the tacrolimus may be adjusted to make sure you are getting the appropriate amount. These adjustments will be made based on the levels of tacrolimus measured in your blood. Adjustments may be made even if you are in the control group and receiving the placebo just to make sure that neither you nor your doctor can figure out which group you have been assigned to.

## **B2. HOW LONG WILL I BE IN THE PROJECT?**

You will be in this research study for about 32 weeks – 30 weeks enrolled in the study, plus about 2 weeks to complete screening procedures. You will take the study drug for 12 weeks.

#### **B3. CAN I STOP BEING IN THE PROJECT?**

You are free to withdraw from the project at any time. If you leave, your regular medical care will not change. If you are thinking about leaving, please tell the research doctor.

- The research doctor can tell you about the effects of stopping, and you and the research doctor can talk about what follow-up care would help you the most.
- You might be asked to come back for one more visit to check your health.
- You might be asked to return your research drug containers.

The research doctor may take you out of this project at any time. This would happen if:

- They think it is in your best interest.
- You do not follow the project rules.
- The whole project is stopped.

If this happens, the research doctor will tell you.

#### **B4. ARE THERE ANY SPECIAL INSTRUCTIONS WHILE I AM IN THE PROJECT?**

You should not eat or drink grapefruit products or take medications called CYP3A inducers or CYP3A inhibitors while on study medication. A list of these medications will be provided to you.

**Informed Consent for Research** 


IRB Protocol Number: PRO00027931

IRB Approval Period: 9/25/2018 - 2/26/2019

## **EFFECTIVE**

9/25/2018

MCW/FH IRB

## C1. WHAT HEALTH RISKS OR PROBLEMS CAN I EXPECT FROM THE PROJECT?

There are risks to taking part in any research project. There is a risk that you may get a drug combination that does not help your condition or may make it worse. There also may be problems (side effects) we do not know about yet, from the drug itself, or how it combines with other drugs you are taking. If we learn about new important side effects, we will tell you.

We watch everyone in the project for problems (side effects). You need to tell the research doctor or a member of the research team immediately if you experience any problems, side effects, or changes in your health.

#### **C2. RISKS OF TACROLIMUS**

The research drug itself may cause problems (side effects). Side effects may be mild or very serious. Some can last a long time or never go away. Many go away soon after you stop taking the drug. Drugs can affect individuals in different ways.

The side effects that other people have experienced so far with the tacrolimus are:

- Kidney injury: patients may develop a rise in serum creatinine (a marker of kidney function), which is usually reversible when decreasing or discontinuing the drug. Chronic kidney damage is rarely seen in patients on short courses of therapy.
- Hypertension: tacrolimus may raise the blood pressure.
- Neurological side effects: Tremors are a common side effects of tacrolimus, and are usually temporary, even without dose adjustment. Rarely, patients may develop headaches. Studies have shown mild tremors in up to 20% of patients and headaches in about 5%. Seizures were previously reported, but they are usually seen with intravenous administration of the drug and patients with previous history of seizures will be excluded from the study.
- Metabolic abnormalities: Tacrolimus may cause high blood sugar, but no severe cases have been reported.
- Rare side effects: loss of appetite, nausea, vomiting, diarrhea, and abdominal discomfort. Increased liver enzymes are reversible with dose reduction or drug discontinuation.
- Infections: there is a theoretical risk of infections in patients on immunosuppressants. Tacrolimus may predispose the patients to infection with pneumocystis jiroveci, a rare type of pneumonia or lung infection.

#### C3. OTHER RISKS OF THIS RESEARCH PROJECT

Other procedures and medications that are part of the research also involve some risks:

- Vedolizumab Most common adverse reactions: nose, mouth, and throat irritation; headache; joint aches; nausea; fever; upper respiratory tract infection; fatigue; cough; bronchitis; influenza; back pain; rash; itching; sinusitis; and pain in extremities.
- PML Both vedolizumab and tacrolimus have warnings in the label for the risk of a rare infection of the brain, called progressive multifocal leukoencephalopathy

#### **Informed Consent for Research**


IRB Protocol Number: PRO00027931

IRB Approval Period: 9/25/2018 - 2/26/2019

#### **EFFECTIVE**

9/25/2018

MCW/FH IRB

(PML). There have been some potential reports of PML associated with immunosuppressant drugs including tacrolimus. There is also a potential risk with vedolizumab, although to date, no cases have been reported that are directly attributed to vedolizumab. Patients will be monitored for any new onset, or worsening, of neurological signs and symptoms, including the typical signs and symptoms associated with PML that are diverse, progress over days to weeks, and include progressive weakness on one side of the body or clumsiness of limbs, disturbance of vision, and changes in thinking, memory, and orientation leading to confusion and personality changes. Since the progression of deficits usually leads to death or severe disability over weeks or

months, the study drug(s) will be stopped immediately if PML is suspected, and the patient will be referred to a neurologist.

- Vaccines You should not receive live vaccines while you are taking tacrolimus.
   The people you live with should also not receive live vaccines. If you or someone you live with needs a vaccine during the course of a study, please talk to a member of the study team.
- Interactions with other medications, herbals, and food Foods (such as grapefruit juice) and medications, including herbal remedies can change the way your body processes the study drugs. A member of the study team will talk to you about your current medications and you should tell someone on the study team before you start any new medications during the study.
- Blood draw The side effects you might experience from giving a blood sample
  for this study include possible discomfort and bruising at the needle entry site. Rare
  complications from any venipuncture (drawing blood from a vein) include fainting, arterial
  puncture, nerve injury, infection, and blood clot. Precautions will be taken to ensure your
  safety and minimize discomfort. The person drawing your blood will observe you for side
  effects.
- Flexible sigmoidoscopy discomforts and risks associated with a sigmoidoscopy include: Heavy or ongoing bleeding from biopsy or removal of polyp; cramping, pain, and abdominal bloating; Peritonitis (inflammation of the lining of the abdominal cavity); Perforation (a hole) of the intestinal wall. Surgery may be needed if a perforation occurs; Nausea, vomiting, bloating, or rectal irritation caused by the bowel cleanse prep; medication side effects, like drowsiness following sedative or pain medication if given; or an allergy to the anesthesia.
- Biopsy biopsy risks include: persistent bleeding at the site of the biopsy; pain; infection. Biopsy results can identify abnormalities and even cancer of the intestine you did not know about.

## **C4. REPRODUCTIVE RISKS**

#### Risks to women who could become pregnant

The drug in this project might affect a baby, before or after the baby is born. We do not know if the drug causes harm to a baby, so we do not want anyone who might be pregnant to enter the project. You should not become pregnant or nurse a baby while in this project. You must tell the research doctor right away if you think you are pregnant. You will be asked to have a pregnancy test to be sure you are not pregnant at the start of the project and periodically during the study.

You may not donate eggs during your participation in the project.

#### **Informed Consent for Research**


IRB Protocol Number: PRO00027931

IRB Approval Period: 9/25/2018 - 2/26/2019

## **EFFECTIVE**

9/25/2018

MCW/FH IRB

If you become pregnant during the project, you will be dropped from participation for safety reasons. If you become pregnant while you are taking this experimental drug, we ask that you inform the research doctor immediately. The research doctor will ask you for written permission to obtain information from you or your obstetrician on your pregnancy and the health of the baby.

## Risks of fathering a child

You should not father a baby while taking part in this project because it is unknown if the drug could affect a baby. If your partner is able to become pregnant, one or both of you must use some form of effective birth control. You must tell the research doctor right away if you think your partner is pregnant.

## Birth control methods for all subjects

Check with the research doctor about the birth control methods needed for this project and how long to use them. Some methods might not be good enough for this project. If you are having sex that could lead to pregnancy, you should use birth control while you are in this project. This may include:

- Not having vaginal sex (abstinence)
- Taking birth control pills orally
- Having birth control shots or patches such as Depo-Provera
- Surgical sterilization (hysterectomy or tubal ligation)
- Use of an intrauterine device (IUD)
- Use of diaphragm with contraceptive jelly
- Use of condoms with contraceptive foam
- Use of diaphragm with condoms ("double barrier")
- Limiting sexual activity to a male partner who has had a vasectomy

If you are not surgically sterile or abstinent, you should use 2 methods of contraception. You should continue using birth control for 4 weeks after stopping the study drug.

## C5. ARE THERE ANY BENEFITS TO TAKING PART IN THE PROJECT?

We don't know if this study will help you. Your condition may get better but it could stay the same or even get worse. We hope the information from this study will help us develop better treatments for ulcerative colitis.

#### D1. ARE THERE ANY COSTS TO BEING IN THE PROJECT?

Most of the medical care that you will receive in this study is considered routine care for your condition and would be recommended whether you join the study or not. Costs for routine care will be billed to you or your insurance carrier.

Activities / costs that are part of the study will not be billed to you or your insurance company. These are:

- Flexible sigmoidoscopy / biopsy
- Urine pregnancy test
- Tacrolimus level
- Magnesium level
- Phosphorus level

**Informed Consent for Research** 


IRB Protocol Number: PRO00027931

IRB Approval Period: 9/25/2018 - 2/26/2019

**EFFECTIVE** 

9/25/2018

MCW/FH IRB

- Tacrolimus or placebo
- Magnesium (if needed)
- Phosphorus
- CBC
- Comprehensive metabolic panel done at times other than screening, week 6, and week
   14
- Fecal calprotectin

Some insurers will not pay for drugs, tests or hospitalization that are part of research studies, so check with your insurer before you join this study. If you have questions regarding study costs, please contact Dr. Yarur.

If you participate in this research, the costs of any necessary emergency medical treatment in the event of a research-related injury will be billed to you or your health insurance.

## D2. WILL I BE PAID FOR PARTICIPATING IN THE PROJECT?

You will receive \$250 for each week you are in the study, for 14 weeks. This totals \$3500. This is to compensate you for time spent on study visits and lab draws, including mileage / travel. If you do not complete 14 weeks of the study, your payments will be prorated by week. To pay you, we need your social security number. Any payment may be reportable as income on your taxes.

#### D3. WHAT OTHER HEALTHCARE CHOICES DO I HAVE?

You do not have to join this project. You are free to say yes or no. If you do not join this project, your research doctor can discuss other healthcare choices with you.

Your other choices may include:

- Not participating in any research and continuing your routine care
- Joining a different research project
- The procedure or drug offered to you may also be available without being in any research project.

The research doctor can explain both the possible benefits and the risks of other options that are available to you.

## D4. WILL I BE GIVEN NEW INFORMATION ABOUT THE PROJECT?

If we learn any important new information about the drugs that might change your mind about being in the project, we will tell you about it right away. You can then decide if you want to stay in the project.

Clinically relevant results, including individual results, will be disclosed to you, when the study is done.

#### **Informed Consent for Research**


IRB Protocol Number: PRO00027931

IRB Approval Period: 9/25/2018 - 2/26/2019

#### **EFFECTIVE**

9/25/2018

MCW/FH IRB

## D5. WHAT HAPPENS IF I AM INJURED BECAUSE I TOOK PART IN THE PROJECT?

Emergency medical treatment for injuries directly related to your participation in this research project will be provided to you. You or your health insurance will be billed for the costs of this emergency treatment. MCW will decide on a case by case basis if they will reimburse you or your insurer for emergency treatment costs. If your research-related injury requires medical care beyond this emergency treatment, you or your insurer will be responsible for the costs of this follow-up care.

At this time, there is no plan for any additional financial payments.

If you believe that you have been injured because of your participation in this project, contact the research doctors right away. Contact information: 414-805-7128 (study team)

Nothing in this consent form affects any legal rights you may have nor does it release the investigator, the sponsor, the institution, or its agents from liability for negligence.

## D6. WHO CAN ANSWER MY QUESTIONS ABOUT THE PROJECT?

- If you have more questions about this project at any time, you can call Dr. Yarur at 414-805-6858.
- If you have questions about your rights as a research participant, want to report any problems or complaints, or offer input, you can call the MCW/Froedtert Hospital Research Subject Advocate at 414-955-8844.

## E. PERMISSION TO COLLECT, USE AND SHARE HEALTH INFORMATION

## E1. What health information will be collected and used for this project?

To be in this research project, the research team needs your permission to access, collect and use some of your health information. If you say no, you cannot be in the project. This information may come from questions we ask, forms we ask you to fill out, or your medical record, as described below. We will only collect and use information needed for the project.

The protected health information (PHI) originates from services you will or have received at one or more of the following locations: the Medical College of Wisconsin (MCW); BloodCenter of Wisconsin (BCW); Children's Hospital of Wisconsin (CHW); any Froedtert Health Affiliate-Froedtert Memorial Lutheran Hospital (FMLH), Inc.; Community Memorial Hospital (CMH) Menomonee Falls, Inc.; St. Joseph's Community Hospital (SJH) West Bend, Inc.; Froedtert & The Medical College of Wisconsin Community Physicians Clinics, Inc. (FMCWCP); the West Bend Surgery Center, LLC; and the Froedtert Surgery Center, LLC.

#### The health information to be collected and used for this project is:

- ⇒ Your medical record as it relates to your ulcerative colitis treatment and diagnosis
- ⇒ Your medical record relating to your care in this study

**Informed Consent for Research** 


IRB Protocol Number: PRO00027931

IRB Approval Period: 9/25/2018 - 2/26/2019

**EFFECTIVE** 

9/25/2018

MCW/FH IRB

## E2. Who will see the health information collected for this project?

The only MCW/Froedtert Hospital employees allowed to handle your health information are those on the research team, those on the Institutional Review Board (IRB) and those who check on the research activities to make sure the hospital's rules are followed.

If the costs of any necessary emergency medical treatment in the event of a research-related injury are billed to your health insurance, your health information may need to be disclosed to the insurer for billing purposes.

Because this project involves the use of drugs and/or devices, the FDA also has the right to inspect all project records.

We may record your research information, including results of tests and procedures done for research, in your Froedtert Hospital and/or Medical College of Wisconsin medical record. As a result, this research information may be seen by people allowed to see your medical records for healthcare operations or treatment, by those you allow to see your medical records by giving written permission, and by others when required by law.

We will not use your personal health information for a different project without your permission or the permission of a hospital research review board (IRB). Once all personal identification is removed from your health information the information may be used for future research or distributed to another investigator for future research without additional informed consent from you or your legally authorized representative. The information might also be used or released for other purposes without asking you. Results of the project may be presented in public talks or written articles, but no information will be presented that identifies you.

#### E3. What are the risks of sharing this health information?

One risk of taking part in a research project is that more people will handle your personal health information collected for this project. The research team will make every effort to protect the information and keep it confidential, but it is possible that an unauthorized person might see it. Depending on the kind of information being collected, it might be used in a way that could embarrass you or affect your ability to get insurance. If you have questions, you can talk to the research doctor about whether this could apply to you.

## E4. How long will you keep the health information for this project?

If you sign this form, we plan to keep your information for 10 years after the research project ends, for paper data collected, and indefinitely for electronic data, in case we need to check it again for this project.

# E5. Can I cancel my permission to share this health information?

If you change your mind later and do not want us to collect or share your health information, you need to send a letter to Dr. Yarur at Medical College of Wisconsin, Division Gastroenterology and Hepatology, 8701 Watertown Plank Road, Milwaukee WI 53226. The letter must say that you have changed your mind and do not want the researcher to collect and share your health

Medical College of Wisconsin & Froedtert Hospital **Informed Consent for Research** 


IRB Protocol Number: PRO00027931

IRB Approval Period: 9/25/2018 - 2/26/2019

**EFFECTIVE** 

9/25/2018

MCW/FH IRB

information. At that time, we may decide that you cannot continue to be part of the project. We may still use the information we have already collected.

## E6. Access to records

If you join this project, you will be given one of two treatments without knowing exactly which one (a "blinded" project). If you ask to see your health records during this "blinded" project, the research team cannot tell you which drug you are being given. This is because the research team also remains "blinded" about which drug the sponsor has randomly assigned to you. You would have to wait until the time given below. We cannot do the project unless you agree. However, if the blinded information is needed to treat you, it will be provided to the research doctor.

- What are the blinded options? You will get one of these drugs/interventions: Vedolizumab and Tacrolimus or Vedolizumab alone
- When can you find out which drug you were given? You can find out 30 weeks after you start the study.

## F1. FOR MORE INFORMATION ABOUT THE PROJECT

A description of this clinical trial will be available on http://www.ClinicalTrials.gov as required by U.S. Law. This Web site will not include information that can identify you. At most, the Web site will include a summary of the results. You can search this Web site at any time.

You can look up this project by referring to the ClinicalTrials.gov number NCT02954159 or by asking the research team for a printed copy.

**Informed Consent for Research** 


IRB Protocol Number: PRO00027931

IRB Approval Period: 9/25/2018 - 2/26/2019

**EFFECTIVE** 

9/25/2018

MCW/FH IRB

#### **CONSENT TO PARTICIPATE**

## By signing my name below, I confirm the following:

- I have read (or had read to me) this entire consent document, including Attachment 1. All of my questions have been answered to my satisfaction.
- The project's purpose, procedures, risks and possible benefits have been explained to me.
- I agree to let the research team use and share the health information and other information gathered for this project.
- I voluntarily agree to participate in this research project. I agree to follow the procedures as directed. I have been told that I can stop at any time.

**IMPORTANT:** You will receive a signed and dated copy of this consent form. Please keep it where you can find it easily. It will help you remember what we discussed today.

| Subject's Name please print | Subject's Signature | Date OR Date/Time |
|---|---|---|
| Name of Witness (if applicable) please print (for short form consent process, or consent of blind or illiterate subject) | Signature of Witness | Date |
| | Signature of person discussing/obtaining consent | Date |
| Name of Principal Investigator please print I participated in consent process I acknowledge enrollment of this subject into the project | Signature of Principal<br>Investigator | Date |

Attachment 1 – Details of project schedule and procedures

**Informed Consent for Research** 


IRB Protocol Number: PRO00027931

IRB Approval Period: 9/25/2018 - 2/26/2019

**EFFECTIVE** 

9/25/2018

MCW/FH IRB

# **Schedule of Events**

| | Pre-<br>treatment | Treatment | | | | | | Follow<br>Up | |
|---|---|---|---|---|---|---|---|---|---|
| Schedule of<br>events | Screening | Week<br>0 | Week<br>2 | Week<br>6 | Week<br>8 | Week<br>12 | Week<br>14 | When needed | Week<br>30 |
| Informed<br>Consent | <u>~</u> | | | | | | | | |
| Begin tacrolimus | | <b>✓</b> | | | | | | | |
| Begin<br>vedolizumab | | <b>V</b> | | | | | | | |
| Stop tacrolimus | | | | | | <u>~</u> | | | |
| Prior<br>medications | V | | | | | | | | |
| Concomitant<br>medications | V | | V | V | V | | ~ | | V |
| Demographics | ~ | | | | | | | | |
| Smoking status | ~ | | | | | | <b>/</b> | | |
| Medical/surgical history | V | | | | | | | | |
| Vitals signs | ~ | <b>✓</b> | <u>~</u> | <u>~</u> | <u>~</u> | | <b>✓</b> | <u>~</u> | <b>/</b> 2 |
| Body mass (Kgs) | ~ | <b>✓</b> | | | | | | | |
| Urine pregnancy test (women) | <u>~</u> | <u> </u> | <u>~</u> | <u>~</u> | | | <b>✓</b> | | |
| Adverse events assessment | | | <u>~</u> | <u>~</u> | <u>~</u> | <u>~</u> | <u>~</u> | <u>~</u> | <u>~</u> |

## **Informed Consent for Research**

Clinical Interventions template - Version: March 30, 2018 IRB Protocol Number: PRO00027931

IRB Approval Period: 9/25/2018 - 2/26/2019

# **EFFECTIVE**

9/25/2018

MCW/FH IRB

| Mayo partial score | <u>~</u> | <u>~</u> | <u>~</u> | <u> </u> | <u>~</u> | <u>~</u> | | <b>✓</b> 2 |
|---|---|---|---|---|---|---|---|---|
| Colonoscopy or sigmoidoscopy | <u>~</u> | | | <u>~</u> | | | • | <b>✓</b> 2 |
| Endoscopic<br>Mayo UC score | <u>~</u> | | | <u>~</u> | | | | <b>✓</b> 2 |
| UCDAI | <b>✓</b> | <u>~</u> | <u>~</u> | <u>~</u> | <u>~</u> | <u>~</u> | | <b>✓</b> 2 |
| CRP | ~ | ~ | | ~ | | ~ | | <b>√</b> 2 |
| C. diff / stool culture | V | | | | | | | |
| Fecal calprotectin | | ~ | | ~ | | <u>~</u> | | <b>✓</b> 2 |
| Comprehensive<br>Metabolic panel | V | ~ | <u>~</u> | ~ | <u>~</u> | ~ | <u>~</u> | <b>/</b> 2 |
| Serum<br>magnesium | V | ~ | <u>~</u> | <u>~</u> | <u>~</u> | <u>~</u> | <u>~</u> | |
| Serum<br>phosphorus | V | ~ | <u>~</u> | <u>~</u> | <u>~</u> | <u>~</u> | <u>~</u> | |
| Tacrolimus level | | <u>~</u> | <u>~</u> | <u>~</u> | <u>~</u> | <u>~</u> | <u>~</u> | |
| Complete blood count | V | ~ | | ~ | | ~ | | <b>/</b> 2 |
| Development of Clostridium Difficile infection? | | | V | ~ | V | • | • | V |
| Discontinuation of therapy? | | | ~ | ~ | ~ | ~ | • | ~ |
| Assessment of Colectomy | | | ~ | ~ | ~ | ~ | | ~ |

Medical College of Wisconsin & Froedtert Hospital **Informed Consent for Research** 


IRB Protocol Number: PRO00027931

IRB Approval Period: 9/25/2018 - 2/26/2019

**EFFECTIVE** 

9/25/2018

MCW/FH IRB

(1) "when needed" lab draws will be done to follow-up labs and adjust the drug if needed. They will be performed before the fourth or fifth dose after a change of tacrolimus dose. Therapeutic drug monitoring: patients will be tested for tacrolimus and serum electrolytes (Na, K, Cl, phosphorus, creatinine, blood urea, magnesium)

(2) Only if performed as a standard of care.